CLINICAL TRIAL: NCT06335342
Title: Radiotherapy Treatments for Neoplasms in the Head and Neck Region
Status: Recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: IEO 0726
Record Dates: First submitted 2024-03-22; First posted 2024-03-28 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-03

CONDITIONS: Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Radiotherapy to head and neck region: Patients treated at European Institute of Oncology with radiotherapy to head and neck region

SUMMARY:
The aim of this study is the evaluation of clinical and dosimetric aspects, tolerance, and effectiveness of radiotherapy treatments in the head and neck region.

Eligible patients undergoing radiotherapy for primary or secondary neoplasms localized in the head and neck anatomical region.

DETAILED DESCRIPTION:
Approximately 60% of patients with neoplasms receive radiotherapy as part of their oncological treatment.

Various primary tumors as well as metastases of various origins can be localized in the head and neck anatomical region. Patients with such neoplastic localizations will therefore receive radiotherapy treatment possibly associated with other systemic or surgical treatments.

Treatment choice is usually established following multidisciplinary discussions, based on disease characteristics and stage, concurrent pathologies and pharmacological treatments, patient preferences, and functional aspects.

The collection of data related to radiotherapy plays a crucial role in understanding various clinical aspects of the treatment itself. The availability of data from an increasing number of patients will allow the identification of clinical situations or technical parameters of radiotherapy correlated with treatment tolerance and effectiveness, aiming to identify the best treatment for these oncological pathologies.

This project aims to collect data related to radiotherapy treatments for primary or secondary neoplasms of the head and neck region for scientific dissemination with the goal of establishing the basis for evaluating achieved results over time, and deriving from these elements useful for guiding the most effective treatment strategies and appropriate operational protocols.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with radiotherapy for curative, palliative, neo-adjuvant, and adjuvant purposes in the head and neck region include those with:

  * Primary bone tumors,
  * Primary soft tissue tumors,
  * Primary tumors of the cardio-circulatory system,
  * Primary tumors of the lymphatic system,
  * Primary tumors of the nervous system and skin,
  * Secondary metastases from various origins localized in that district.
* Signed informed consent

Exclusion Criteria:

• Radiotherapy in districts other than the head and neck region

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated at European Institute of Oncology with radiotherapy for curative, palliative, neo-adjuvant, and adjuvant purposes in the head and neck region
Sampling Method: Non-Probability Sample
Enrollment: 4050 (Estimated)
Dates: Start 2018-02-22 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 5 years
  Number of patients death
Disease free survival | 5 years
  Number of oncological event (local recurrence, distant metastasis, other primary tumor)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Alicja Jereczek, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy